CLINICAL TRIAL: NCT03802500
Title: Early Electromyographic Evaluation of the ICU-acquired Weakness in Septic Shock Patients Ventilated Longer Than 72 Hours: Neurophysiological Study
Brief Title: Neurophysiological Diagnosis for ICU Septic Shock Patients
Acronym: EDX
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Universitaire Vaudois (Other)
Responsible Party: Principal Investigator, CAROLINE ATTWELL, Mrs, Centre Hospitalier Universitaire Vaudois
Other Study IDs: NRA-01
Record Dates: First submitted 2018-12-12; First posted 2019-01-14 (Actual); Last update posted 2019-10-04 (Actual); Status verified 2019-10

CONDITIONS: ICU Acquired Weakness
MeSH Terms: interventions — Nerve Conduction Studies

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Diagnostic Test: Nerve conduction study — Physical examination of muscle strength is conducted using the Medical Research Council (MRC) scale in 6 muscles bilaterally.
  Patients with an MRC score of less than 48 of 60 are diagnosed with critical illness polyneuromyopathy (CIPNM).
  The evaluation is completed by a routine neurological examination. In patients meeting the inclusion criteria, the screening Peroneal nerve test (PENT test) is performed on the day of study enrollment and subsequently in 1 week intervals until pathologic findings are detected or patient is discharged from the ICU.
  PENT measures the peroneal nerve Compound muscle action potential (CMAP) amplitude in one leg. If the PENT is normal, the contra-lateral peroneal nerve is measured. An abnormal condition is identified if the peroneal nerve CMAP amplitude is reduced below the normal limits of the participating centre in at least one leg. In Lausanne, the abnormal response is < 2,5 mV.
  Other Names: Peroneal nerve test (PENT test)

SUMMARY:
Patients hospitalized in the Intensive Care Unit (ICU) are at risk for developing severe disabilities, physical or cognitive. In particular, ICU-acquired weakness is frequent. The causes of this weakness are multiple and the physiopathology is still not fully understood. Immobilization in bed and sepsis are known risk factors.

ICU-acquired weakness has been associated with prolonged mechanical ventilation duration, and increased in ICU and hospital length of stay. It has also been associated with significant decrease in functional capacity and with higher mortality. An early screening using a specific diagnostic protocol could help improving the management of patients suffering from ICU acquired weakness.

The aim of this study is to early detect ICU acquired weakness in patients suffering from septic shock and ventilated for more than 72 hours.

ELIGIBILITY:
Inclusion Criteria:

• Patients admitted to the ICU with a septic shock and ventilated for more than 72 hours.

Exclusion Criteria:

* Hospitalization for more than 7 days before intubation.
* Functional disability at admission of ≥4 (Requires constant nursing care and attention, bedridden, incontinent) in the Modified Rankin Scale.
* Lower limb disorders precluding nerve conduction studies (NCV) and electromyography (EMG), such as clinical edema of the lower limbs, or fractures, amputation, and plaster casts of the lower limbs.
* Evidence of altered neuromuscular transmission at repetitive stimulation test either caused by neuromuscular blocking agents or disease.
* Burn patients admitted to ICU.
* Patient requesting withdrawal of therapies.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted to the ICU with a septic shock and ventilated for more than 72 hours.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2019-01-23 (Actual); Primary Completion 2019-10-31 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
Presence of ICU-acquired weakness in septic shock patients ventilated for more than 72 hours. | 72 hours
  Medical Research Council strength scale

SECONDARY OUTCOMES:
ICU length of stay | Up to 6 months
Hospital length of stay | Up to 6 months
Discharge destination | At discharge from hospital, up to 6 months
Length of ventilatory support | At extubation, up to 6 months
Extubation failure rate | up to 72 hours, after first extubation
  Patients requiring reintubation 72 hours after failed first extubation
Time elapsed between endotracheal intubation and first out-of-bed mobilization | up to 6 months, at first out-of-bed mobilization

CONTACTS AND LOCATIONS:
Overall Officials: Karin Diserens, PD-MER, Study Director — NRA Unit. CHUV.
Locations (1):
- CHUV, Lausanne, Canton of Vaud, Switzerland

IPD SHARING:
Plan to Share IPD: No